CLINICAL TRIAL: NCT06205836
Title: Evaluating a Surgical-Sparing Approach Using Cemiplimab With or Without Fianlimab to Treat Older Patients With Localized or Locally Advanced MSI-H Colorectal Cancer
Brief Title: Cemiplimab With or Without Fianlimab to Treat Older Patients With Localized or Locally Advanced MSI-H Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J23155; IRB00415816 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Cemiplimab; Fianlimab; Immunotherapy; Anti-PD-1 therapy; Anti-Lag-3; Adenocarcinoma; Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma; Carcinoma | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A - Cemiplimab (Experimental)
  Interventions: Drug: Cemiplimab
- Cohort B - Cemiplimab with Fianlimab (Experimental)
  Interventions: Drug: Cemiplimab; Drug: Fianlimab
- Cohort C - Cemiplimab (Experimental)
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Patients will receive cemiplimab (350 mg administered IV) on Day 1 of each 21 day cycle for a total of 4 cycles of treatment.
  Other Names: REGN2810, LIBTAYO
Drug: Fianlimab — Patients will receive fianlimab (1600 mg administered IV) on Day 1 of each 21 day cycle for a total of 4 cycles of treatment.
  Other Names: REGN3767
  Arms: Cohort B - Cemiplimab with Fianlimab

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of cemiplimab and the combination of cemiplimab/fianlimab in microsatellite unstable localized or locally advanced colorectal cancer diagnosed in patients age 70 or greater or in patients age 18 or greater considered poor candidates for surgery.

ELIGIBILITY:
Inclusion Criteria for Cohort A and B:

* Age ≥70 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
* Have histologically proven localized or locally advanced mismatch repair deficient (dMMR) or microsatellite unstable (MSI-H) colorectal cancer.
* Must not have received any prior systemic treatment or radiation.
* Must be agreeable to endoscopic, and CT surveillance for a total of 24 months.
* Patient's acceptance to have a tumor biopsy.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests and procedures.
* LVEF assessment with documented LVEF ≥ 45% by either TTE or MUGA (TTE preferred) within 6 months from first study drug administration.
* For both Women and Men, must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Inclusion Criteria for Cohort C:

* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -3.
* Have histologically proven localized or locally advanced mismatch repair deficient (dMMR) or microsatellite unstable (MSI-H) colorectal cancer.
* Patient deemed a poor surgical candidate after evaluation by a surgeon.
* Must not have received any prior systemic treatment or radiation.
* Must be agreeable to endoscopic, and CT surveillance for a total of 24 months.
* Patient's acceptance to have a tumor biopsy.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests and procedures.
* For both Women and Men, must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria for Cohorts A and B:

* Have received an investigational agent or used an investigational device within 28 days of the first dose of study drug.
* Have expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Have had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.).
* History of prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, or anti-Lag-3 antibodies for any reason in the 5 years proceeding their colorectal cancer diagnosis.
* Currently using any chronic systemic steroids.
* Patient has received a live vaccine within 30 days of the first dose of study drug.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active autoimmune disease.
* Any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft.
* Patient has a pulse oximetry of <92% on room air.
* Patient is on supplemental home oxygen.
* Has clinically significant heart disease.
* Cohort B Only: Troponin T (TnT) or troponin I (TnI) > 2x institutional ULN at baseline.
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures.
* Unwilling or unable to follow the study schedule for any reason

Exclusion for Cohort C:

* Have received an investigational agent or used an investigational device within 28 days of the first dose of study drug.
* Have expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Currently using any chronic systemic steroids.
* Patient has received a live vaccine within 30 days of the first dose of study drug.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft.
* Patient is pregnant or breastfeeding.
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures.
* Participation deemed not in the best interest of the patient.
* Unwilling or unable to follow the study schedule for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 6 Months
  Proportion of subjects with either a pathologic complete response (pCR) at the time of surgery OR a clinical complete response (cCR) at 6 months for those subjects who do not undergo surgery. pCR is defined as subjects with no viable tumor cell noted on pathological evaluation of the resection specimen. cCR is defined as an absence of visible disease on CT imaging by RECIST 1.1 and endoscopic evaluation.

SECONDARY OUTCOMES:
Number of participants experiencing grade 3 or above drug-related toxicities requiring treatment discontinuation | 7 Months
  Defined using NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Christenson, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center Johns Hopkins Medical Institution
Locations (1):
- Johns Hopkins SKCCC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No